CLINICAL TRIAL: NCT06619665
Title: A Randomized, Double-blind, 3-Period Crossover Study to Assess the Effects of MK-6552 on Sleep Latency in Sleep Deprived Healthy Participants With Modafinil as a Positive Control
Brief Title: A Study of MK-6552 in Sleep Deprived Healthy Participants (MK-6552-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 6552-003; MK-6552-003 (Other: MSD)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MK-6552-Placebo-Modafinil (Experimental): Participants were treated in period 1 with MK-6552; in period 2 with placebos to Modafinil and MK-6552; and in period 3 with Modafinil; with a 7-day washout between each period.
  Interventions: Drug: MK-6552; Drug: MK-6552 placebo; Drug: Modafinil; Drug: Modafinil placebo
- MK-6552-Modafinil-Placebo (Experimental): Participants were treated in period 1 with MK-6552; in period 2 with Modafinil; and in period 3 with placebos to Modafinil and MK-6552; with a 7-day washout between each period.
  Interventions: Drug: MK-6552; Drug: MK-6552 placebo; Drug: Modafinil; Drug: Modafinil placebo
- Placebo-Modafinil-MK-6552 (Experimental): Participants were treated in period 1 with placebos to Modafinil and MK-6552; in period 2 with Modafinil; and in period 3 with MK-6552; with a 7-day washout between each period.
  Interventions: Drug: MK-6552; Drug: MK-6552 placebo; Drug: Modafinil; Drug: Modafinil placebo
- Placebo-MK-6552-Modafinil (Experimental): Participants were treated in period 1 with placebos to Modafinil and MK-6552; in period 2 with MK-6552; and in period 3 with Modafinil; with a 7-day washout between each period.
  Interventions: Drug: MK-6552; Drug: MK-6552 placebo; Drug: Modafinil; Drug: Modafinil placebo
- Modafinil-MK-6552-Plaebo (Experimental): Participants were treated in period 1 with Modafinil; in period 2 withMK-6552; and in period 3 with placebos to Modafinil and MK-6552; with a 7-day washout between each period.
  Interventions: Drug: MK-6552; Drug: MK-6552 placebo; Drug: Modafinil; Drug: Modafinil placebo
- Modafinil-Plaebo-MK-6552 (Experimental): Participants were treated in period 1 with Modafinil; in period 2 with placebos to Modafinil and MK-6552; and in period 3 with MK-6552; with a 7-day washout between each period.
  Interventions: Drug: MK-6552; Drug: MK-6552 placebo; Drug: Modafinil; Drug: Modafinil placebo

INTERVENTIONS:
Drug: MK-6552 — MK-6552 gelatin coated capsules taken orally two times 8 hours apart
Drug: MK-6552 placebo — MK-6552 placebo gelatin coated capsules taken orally two times 8 hours apart
Drug: Modafinil — Modafinil tablet taken once orally
Drug: Modafinil placebo — Modafinil placebo tablet taken once orally

SUMMARY:
This study examined the safety of the drug MK-6552 and if people tolerated it. It also studied whether MK-6552 works better than placebo for staying awake in sleep deprived healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Criteria include but are not limited to the following:

* Is in good health
* Body Mass Index (BMI) between 18 and 32 kg/m^2, inclusive.

Exclusion Criteria:

Criteria include but are not limited to the following:

* History of or current hypertension,
* Has a history of sleep disorders:

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Participants with an Adverse Event (AE) | Up to Day 30
  Percentage of participants with at least one AE
Participants who discontinued from study due to an AE | Day 1
  Percentage of participants who discontinued from study due to an AE
Maintenance of Wakefulness Test (MWT) for MK-6552 | Postdose time to maximum plasma concentration (Tmax) (at designated timepoints up to 24 hours postdose)
  Sleep latency of MWT for MK-6552 compared with placebo

SECONDARY OUTCOMES:
Area under the concentration=time curve (AUC) for plasma MK-6552 | At designated timepoints up to 24 hours postdose
  AUC for plasma MK-6552 from 0-24 hours postdose
Concentration of plasma MK-6522 at Tmax following morning (AM) dose | Tmax following AM dose (at designated timepoints up to 24 hours postdose)
  Plasma concentration of MK-6552 at Tmax following AM dose
Concentration of plasma MK-6522 at Tmax following afternoon (PM) dose | Tmax following PM dose (at designated timepoints up to 24 hours postdose)
  Plasma concentration of MK-6552 at Tmax following PM dose
Concentration of plasma MK-6552 8 hours (C8h) after first dose | 8 hours
  C8h of plasma MK-6552 after first dose
Concentration of plasma MK-6552 24 hours (C24h) after first dose | 24 hours
  C24h of plasma MK-6552 after first dose
MWT for Modafinil | 2 hours postdose
  Sleep latency of MWT for Modafinil compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - NeuroTrials Research Inc (Site 0001), Atlanta, Georgia
  - Clinilabs (Site 0003), Eatontown, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com